CLINICAL TRIAL: NCT02857530
Title: Efficacy and Safety of Thrombopoietin In Patients With Severe and Very Severe Aplastic Anemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, ZhongHong Shao, head of department of Hematology, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB2013-066-01
Record Dates: First submitted 2016-07-26; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Anemia, Aplastic
MeSH Terms: conditions — Anemia, Aplastic | interventions — Thrombopoietin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhTPO (Experimental): rhTPO injection
  Interventions: Drug: rhTPO
- control (Placebo Comparator): without rhTPO injection
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rhTPO — rhTPO
  Other Names: Recombinant Human Thrombopoietin
  Arms: rhTPO
Drug: placebo — without rhTPO
  Other Names: without Recombinant Human Thrombopoietin
  Arms: control

SUMMARY:
Efficacy and Safety of Recombinant human thrombopoietin in patients with severe aplastic anemia and very severe aplastic anemia, a randomized, double-blind, placebo-controlled, II phase, multi-center clinical research.

DETAILED DESCRIPTION:
rhTPO

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Have severe or very severe aplastic anemia

Exclusion Criteria:

* Have diagnosis of Fanconi anemia
* Have infection not adequately responding to appropriate therapy
* Have Paroxysmal Nocturnal Hemoglobinuria (PNH) clone size in neutrophils of greater than or equal to 50%
* Have creatinine and/or blood urea nitrogen (BUN) ≥2 times the upper limit of normal
* Have serum bilirubin ≥ 1.5 times the upper limit of normal, or ≥4.0 times the upper limit of normal if the patient has been treated with Anti-Thymocytes globulin（ATG） within three weeks of screening.
* Have glutamic-oxaloacetic transaminase （AST） and/or glutamic-pyruvic transaminase （ALT） ≥ 3 times the upper limit of normal
* Are female and are nursing or pregnant or are unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 3 or greater
* Have had other Thrombopoietin (TPO-R) agonists medication in the previous 4 weeks.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Time to platelet transfusion independence in patients at 6 month | 6 month

SECONDARY OUTCOMES:
Time to patients achieve a platelet count 30×10^9/L, 50×10^9/L or100×10^9/L | up to 1year
Overall response rate up to 1 year after Immunosupressive therapy. | up to 1 year
Megakaryocyte, granulocyte and erythrocyte recovery in bone marrow up to 1 year after IST. | up to 1 year
Time to red blood cell/platelet transfusion independence in patients up to 1 year after IST | up to 1 year
Percentage of patients achieve red blood cell/platelet transfusion independence at 3, 6, 9 and 12 months after IST. | up to 1 year
Intervals of red blood cell/platelet transfusion up to 1 year after IST. | up to 1 year
The reticulocyte count of patients up to 1 year after IST. | up to 1 year
Hospitalization days of patients. | up to 1 year
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 1 year
Median hematopoietic response rate up to 1 year after IST. | up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Zonghong Shao, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No